CLINICAL TRIAL: NCT05213442
Title: Liver Status in Psychiatric Inpatients
Acronym: LIVERSPIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital le Vinatier (Other)
Collaborators: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021-A02796-35
Record Dates: First submitted 2022-01-26; First posted 2022-01-28 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Psychiatric Illness
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Intervention Model Description: Monocentric, non randomized, non comparative cross-sectional study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All inpatients in Vinatier psychiatric Hospital (Other): All hospitalized patients can potentially be recruited. They will benefit from the usual clinical and paraclinical examinations as part of their hospitalization diagnostic work-up. For the determination of biological analyses, a blood sample will be taken following inclusion as well as a Fibroscan examination.
  Interventions: Diagnostic Test: To estimate the prevalence rates of liver disease in psychiatric inpatients and to explore factors associated with the existence of liver disease.

INTERVENTIONS:
Diagnostic Test: To estimate the prevalence rates of liver disease in psychiatric inpatients and to explore factors associated with the existence of liver disease. — Patients will receive the usual clinical and paraclinical examinations as part of their hospitalization diagnostic workup. For the biological analyses, a blood sample will be taken following inclusion as well as a Fibroscan examination.
  Data will be collected from the patient, or if necessary from the health care team, using the medical record (interview and/or self-questionnaires).

SUMMARY:
Adults hospitalized in psychiatry have an increased frequency of somatic disorders, in particular various liver diseases (viral hepatitis, non-alcohol related liver steatosis, alcohol related liver disease).

The evaluation of these liver disorders in psychiatric inpatients remains very little explored in France, contributing to the poor overall medical status of psychiatric patients.

The LIVERSPIN study aims to estimate the prevalence rates of liver pathologies in psychiatric inpatients and to explore the factors associated with the existence of a liver pathology

DETAILED DESCRIPTION:
The LIVERSPIN study aims to estimate the prevalence rates of liver disease in psychiatric inpatients and to explore factors associated with the existence of liver disease.

All hospitalized patients can potentially be recruited. They will benefit from the usual clinical and paraclinical examinations as part of their hospitalization diagnostic work-up. For the determination of biological analyses, a blood sample will be taken following inclusion as well as a Fibroscan examination.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years old
* Social insurance
* Current hospitalization in any psychiatric unit of the participating center
* Adult or legal representative who has given written and informed consent to participate in the study. By default, the oral consent of the adult will be obtained (as well as the written consent of the legal representative)
* Information given to the curator(for people under curatorship)

Exclusion Criteria:

* - Clinical state of the patient which do not allow the collection of study data (according to the investigator)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2022-04-06 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
HCV diagnosis | At inclusion
  HCV diagnosis defined by positive HCV antibodies in blood

SECONDARY OUTCOMES:
HBV diagnosis | At inclusion
  HBV diagnosis defined by positive HBsAg in blood
HIV diagnosis | At inclusion
  HIV diagnosis defined by positive anti-HIV1 or anti-HIV2 antibodies in blood
Suspicion of NAFLD | At inclusion
  Suspicion of NAFLD on FIB-4 and the interrogation
Suspicion of alcoholic liver disease | At inclusion
  Suspicion of alcoholic liver disease on FIB-4 and the interrogation

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin ROLLAND, MD, PhD, Principal Investigator — CH LE VINATIER
Locations (1):
- Centre Hospitalier Le Vinatier, Bron, Auvergne-Rhône-Alpes, France

IPD SHARING:
Plan to Share IPD: No